CLINICAL TRIAL: NCT03266198
Title: Fetal Body Composition and Volumes Study
Brief Title: Fetal 3D Study (Fetal Body Composition and Volumes Study)
Status: Completed | Type: Observational
Sponsor: Katherine Grantz (NIH)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Katherine Grantz, Investigator, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Organization: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: 16-CH-N071; NCT02692924 (obsolete NCT alias)
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Fetal Growth Restriction; Fetal Growth Abnormality
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Normal fetal growth is a critical component for a healthy pregnancy and for ensuring the health and well-being of infants throughout childhood and adolescence. One promising area of research suggests that changes in fetal soft tissue may be the earliest changes that occur in pathologic growth. Three-dimensional volume assessments may be used to detect changes in fetal lean mass, fat mass, and organ size that result from pathologic growth earlier than conventional 2D measures. This knowledge may lead to interventions that could minimize or prevent pregnancy and newborn health problems in the future.

DETAILED DESCRIPTION:
The NICHD Fetal Growth Study was a multi-site, prospective cohort study designed to establish a standard for normal fetal growth (velocity) and size for gestational age in the U.S. population. For the singleton study, 2,334 low-risk, non-obese gravidas were recruited from each of 4 self-identified race/ethnicity backgrounds. An additional 468 obese women and 171 dichorionic twin gestations were recruited. After an initial sonogram in the first trimester, women were randomized to serial ultrasonology schedules. Each schedule comprised five additional sonograms for fetal biometry (six in twins) plus additional image and 3D volume acquisition for later analysis.

Ultrasound measurements at each follow-up visit included standard fetal biometrics ((BPD, HC, AC, FL) and the following volumes in the singleton study if they were able to be obtained: 1st trimester: fetus and gestational sac; 2nd and 3rd trimesters: head, cerebellum, face, chest, heart, abdomen, pelvis, arm and thigh. In twins, the volumes collected were 1st trimester: fetus and gestational sac and in the 2nd and 3rd trimesters the thigh. In addition to ultrasound, this study recorded maternal anthropometrics and a brief interview to capture changes in health status, stress and depression, and physical activity at each follow-up visit. Blood draws at baseline and at targeted gestational ages were obtained for the eventual identification of biomarkers indicative of fetal growth were collected. After delivery, neonatal anthropometric measures were assessed, placental biospecimens were collected, and select information about the obstetrical course and newborn status were abstracted from medical charts.

The Fetal 3D Study is being conducted to catalog and perform 2 Dimensional (2D) and 3 Dimensional (3D) measurement of the obstetrical ultrasound images in the existing bank of singleton and twin gestations collected from the NICHD Fetal Growth Studies. The research study aims to understand the relationship between gravid diseases and longitudinal changes in fetal body composition (subcutaneous fat, lean mass) and organ measurements (in singletons) over the course of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women with ultrasound data collected from the NICHD Fetal Growth Studies-Singletons and Twin Gestations

Exclusion Criteria:

* None

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants from the NICHD Fetal Growth Studies-Singletons and Twin Gestations
Sampling Method: Non-Probability Sample
Enrollment: 2809 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Standards for fetal body composition and organ volumes by maternal race/ethnicity | 3 years
  Growth trajectories in singletons and dichorionic twin pregnancies will be created using two- and selected three-dimensional ultrasound measures. Measures in singletons include fetal body composition from 2D abdominal circumference, arm and thigh volumes; cerebellum; adrenal glands; kidneys; liver; pancreas; lungs; first trimester gestational sac, embryo and placenta, using standardized protocols. Measures in twins include 2D abdominal circumference and thigh volumes, and first trimester gestational sac, embryo and placenta.
  Measurements will be performed using stored ultrasound images and 3D volumes that were collected in the NICHD Fetal Growth Studies - Singleton and Twins ClinicalTrials.gov Identifier: NCT00912132 and NCT01369940, respectively. Women were recruited during the first trimester and followed until delivery. Each woman had scheduled ultrasound examinations, one at enrollment and five during follow-up visits (six for twins).
Comparison of fetal 2D and 3D in pregnancies with complications with fetuses in the singleton standard | 3 years
  The study will assess the relationship between gravid diseases and longitudinal changes in fetal body composition (subcutaneous fat and lean body mass) and organ volumes, and compare to those fetuses growing under optimal circumstances (i.e., singleton gestations included in the development of the fetal growth standard.
Investigation of organ volumes (and ratios to fetal weight) and mass (fat) size in association with gravid or neonatal complications, such as kidney to fetal weight in fetal growth restriction, and liver to fetal weight in diabetes, by race/ethnicity | 3 years
Exploration of factors that influence these associations | 3 years
  The study will determine whether potentially modifiable factors including maternal BMI, weight gain, longitudinal changes in maternal body composition, and nutrition and lifestyle factors modifies the relationship between longitudinal changes in fetal body composition (subcutaneous fat and lean body mass) and organ volumes and gravid diseases, and whether they vary by plurality (singleton or twin).
Biomarkers in relation to fetal body composition and 3D volumes | 3 years
  Longitudinal data will compare singleton and twin gestations with respect to maternal biomarkers of fetal growth, well-being and maternal nutritional status using banked biospecimens to determine if the biomarkers ranges established for singletons are applicable to twin gestations.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will generate de-identified data derived from human subjects along with various types of analysis to identify unique points of interest and relationships to relevant associated data such as phenotype and/or social states. All information necessary to interpret the data, such as study protocols, data collection instruments, or survey tools will be clearly documented. Data generated by this project will be shared through the NICHD Data and Specimen Hub (DASH), an NIH-funded/-approved public repository.
Time Frame: Data will be shared at the time of publication or shortly thereafter.
Access Criteria: Any use of this data by a secondary party after submission to the designated repositories must be shared by that party according to the permissions granted by the original consent form of the study participants unless additional permissions are obtained. Secondary parties must adhere to the NIH Human Data Sharing guidelines for broad data sharing and to the limitations for use set forth by the Institutional Certification associated with this project.
URL: https://dash.nichd.nih.gov/

REFERENCES:
- [Derived] Wagner KA, Chen Z, Hinkle SN, Gleason JL, Lee W, Grobman WA, Owen J, Newman RB, Skupski DW, He D, Sherman S, Gore-Langton RE, Zhang C, Grewal J, Grantz KL. Relationship between gestational weight gain with fetal body composition and organ volumes in the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Fetal Dimensional Study: a prospective pregnancy cohort. Am J Clin Nutr. 2025 Feb;121(2):367-375. doi: 10.1016/j.ajcnut.2024.12.007. Epub 2025 Jan 16. PMID 39909708